CLINICAL TRIAL: NCT00004204
Title: A Phase II Study of Temozolomide in the Treatment of Recurrent Malignant Gliomas
Brief Title: Temozolomide in Treating Patients With Recurrent or Progressive Malignant Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067449; CPMC-IRB-8622; SPRI-CPMC-IRB-8622
Record Dates: First submitted 2000-01-21; First posted 2003-07-18 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2006-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Astrocytoma; Oligodendroglioma | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients who have recurrent or progressive malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free survival and response rate of patients with recurrent or progressive malignant glioma treated with temozolomide.
* Determine whether certain categories of malignant gliomas, such as oligodendroglioma, are more sensitive to temozolomide.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients are stratified according to histologic categories (recurrent glioblastoma multiforme [closed to accrual 11/30/01] vs recurrent anaplastic astrocytoma vs recurrent anaplastic oligodendroglioma).

Patients receive oral temozolomide twice daily for 5 consecutive days. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent or progressive malignant glioma of one of the following types:

  * Anaplastic oligodendroglioma or oligoastrocytoma
  * Anaplastic astrocytoma
  * Glioblastoma multiforme (stratum closed to accrual 11/30/01)
* Patients who have failed radiotherapy are eligible
* Measurable disease by CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* SGOT or SGPT less than 3 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2 times ULN (if greater than 2 times ULN then a gamma glutamyl transferase test must be performed)

Renal:

* BUN less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No other serious concurrent infection or other medical illness that would preclude study entry
* No frequent vomiting or partial bowel obstruction
* HIV negative
* No AIDS-related illness
* No other concurrent malignancy except carcinoma in situ of the cervix or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent epoetin alfa

Chemotherapy:

* At least 6 weeks since other prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior radiotherapy (exceptions allowed for recurrent/progressive disease at discretion of primary investigator)

Surgery:

* Recovered from prior surgery

Other:

* No other concurrent investigational agents
* Concurrent anticonvulsant therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Overall Officials: Casilda Balmaceda, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (10):
- United States (10):
  - Stanford University Medical Center, Stanford, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Cancer Center of Albany Medical Center, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Nalitt Institute for Cancer And Blood Related Diseases, Staten Island, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Neurological Clinic, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin